CLINICAL TRIAL: NCT00761566
Title: Double Blind Randomized Controlled Trial of the Effect of Remote Preconditioning on the Exercise Performance of the Elite Swimmers
Brief Title: The Effect of Remote Preconditioning on the Exercise Performance of the Elite Swimmers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Andrew Redington, Head, Heart Centre-Cardiology Division, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 1000012617
Record Dates: First submitted 2008-09-26; First posted 2008-09-29 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: Elite swimmers; Exercise; Preconditioning
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Other: Real preconditioning followed by Sham preconditioning
- 2 (Experimental)
  Interventions: Other: Sham preconditioning followed by Real preconditioning

INTERVENTIONS:
Other: Real preconditioning followed by Sham preconditioning — Subjects in this arm of the study will first receive four 5 minute cycles of upper limb ischemia interspaced with 5 minutes of reperfusion by using a blood-pressure cuff inflated to a pressure of 15 mmHg greater than systolic arterial pressure. The subjects will then cross-over to the other arm of the study and receive four 5 minute cycles of upper limb ischemia interspaced with 5 minutes of reperfusion by using a sham procedure consisting of inflating the blood pressure cuff to 10 mmHg.
  Arms: 1
Other: Sham preconditioning followed by Real preconditioning — Subjects in this arm of the study will first receive four 5 minute cycles of upper limb ischemia interspaced with 5 minutes of reperfusion by using a sham procedure consisting of inflating the blood pressure cuff to 10 mmHg. They will then cross-over to the other arm of the study and receive four 5 minute cycles of upper limb ischemia interspaced with 5 minutes of reperfusion by using a blood-pressure cuff inflated to a pressure of 15 mmHg greater than systolic arterial pressure.
  Arms: 2

SUMMARY:
In this study, we will test the hypothesis that preconditioning highly trained swimmers using skeletal muscle ischemia as the stimulus will improve exercise performance assessment.

DETAILED DESCRIPTION:
The main purpose of this study is to determine if it is possible to precondition competitive swimmers and improve their exercise performance to provide further insight into the physiological mechanisms through which preconditioning may function. With four 5 minute inflation cycles of a blood-pressure cuff, we will induce skeletal muscle ischemia which is known to be a powerful method of preconditioning. Each swimmer will be blinded to the expected effect and randomly assigned to real preconditioning versus the sham intervention which will consist of four 5 minute cycles of blood pressure cuff inflation to 10mmHg. During a subsequent training session, the subjects will receive the intervention they have not received during the previous test session. Therefore, each subject will be part of both study groups and will serve as their own control. To evaluate the exercise performance, the subjects will perform an incremental swimming test protocol based on methods developed and reported by a member our research team. Swimming velocity, blood lactate level, heart rate, breathing frequency, dyspnoea and oxygen saturation will be measured during incremental exercise. Finally, we would like to determine the preconditioning effect of regular exercise training in an animal model.

Exercise performance is thought to be limited by skeletal, cardiac and respiratory muscle fatigue associated with episodes of exercise induced arterial hypoxemia. Preconditioning is defined as a period of brief lack of oxygen or ischemia in a tissue that protects the heart or any other organ from another sustained episode of ischemia. Preconditioning is believed to improve exercise performance by protecting the skeletal, cardiac and respiratory muscles against decreased oxygen and by-products of anaerobic metabolism that may limit an individual's exercise performance. Elite athletes, such as highly trained swimmers, may provide the research team with the opportunity to evaluate the effect of preconditioning during local tissue hypoxia and anaerobic metabolic by-products in healthy adolescents, which is otherwise not possible. With this study, we will show if it is possible to precondition competitive swimmers and improve their exercise performance using ischemia of the limb as a preconditioning stimulus.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female athlete volunteers
* Post-pubescent swimmers between the ages of 13 and 22 years (or healthy non-athletes (for the "equipment control" group and for the control arm for the animal model section)
* Members of competitive swimming teams
* Have achieved a swimming performance time within 5% of national qualification standards

Exclusion Criteria:

* Illness, surgery, or medical intervention within the last 48 hours
* Diabetes mellitus

Ages: 13 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Improvement in the peak velocity in the preconditioning subjects. | 2 weeks

SECONDARY OUTCOMES:
Breathing frequency. | 2 weeks
Blood lactate. | 2 weeks
Improvement in critical speed. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Redington, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Toronto Swim Club, University of Toronto Athletic Centre, Toronto, Ontario, Canada